CLINICAL TRIAL: NCT00843076
Title: Impact of the Hepatitis C Virus Variability on Liver Steatosis
Brief Title: Impact of Hepatitis C Virus Variability on Steatosis
Acronym: Viro-steatosis
Status: Terminated | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital, Tours, University Hospital, Tours
Other Study IDs: AORT08-PR/VIRO-Stéatose
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy
  Blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic infection by the hepatitis C virus (HCV) is a common cause of liver disease, which may progress to cirrhosis and eventually liver cancer. The therapeutic indication will depend mainly on the importance of liver damage (fibrosis), which can be assessed by physical techniques, blood tests and a liver biopsy. The overall objectives of the project are to understand how HCV variability may influence the severity of steatosis (accumulation of fat in the liver), studying 30 patients chronically infected with HCV (half of these patients infected by HCV genotype 3, versus the other half infected by HCV of another genotype). A small portion of the biopsy performed for the routine pathology examination will be placed in special fixation buffer for electron microscopy (EM). Counting and measuring the size of lipid droplets present in the liver by EM will be used to precisely quantify and characterize the liver steatosis. A blood sample of patients will also be collected to sequence the viral genome present in the patient and identify the amino acids involved in an increase in intracellular accumulation of lipid droplets. This work should clarify the impact of the viral variability in the severity of steatosis. Ultimately, the identification of viral sequences responsible for an increase of this phenomenon could be crucial for understanding the mechanisms involved in the steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C, naive of an antiviral treatment or after relapse or non-response for an antiviral treatment stopped for more than 1 year
* Liver biopsy necessary for the care of the patient
* Signature of informed consent

Exclusion Criteria:

* Patients for which the liver biopsy is estimated ≤ 18 mm, so a portion of 3 mm could not be devoted for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROINGEARD, Study Director — INSERM ERI 19
Locations (6):
- France (6):
  - CH de Blois, Blois
  - CH de Bourges, Bourges
  - CH de Châteauroux, Châteauroux
  - CH de Dreux, Dreux
  - CHR Orléans, Orléans
  - CHRU de Tours, Tours